CLINICAL TRIAL: NCT03349606
Title: Imaging of Cortical Dopamine Transmission in Cocaine Dependence
Brief Title: Cocaine Use Disorder and Cortical Dopamine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajesh Narendran, Visiting Professor in Radiology, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO10030625; R01DA026472 (NIH); PRO14080588 (Other: University of Pittsburgh)
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Dextroamphetamine

STUDY DESIGN:
Intervention Model Description: [C-11]FLB 457 d-amphetamine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cocaine dependence (Experimental): [C-11]FLB 457 PET at baseline and post d-amphetamine
  Interventions: Drug: d-amphetamine; Radiation: [C-11]FLB 457
- Controls (Experimental): [C-11]FLB 457 PET at baseline and post d-amphetamine
  Interventions: Drug: d-amphetamine; Radiation: [C-11]FLB 457

INTERVENTIONS:
Drug: d-amphetamine — oral d- amphetamine 0.5 mg/kg is used to stimulate dopamine release in the brain
Radiation: [C-11]FLB 457 — PET radiotracer

SUMMARY:
The goal of this study is to use [C-11]FLB 457 and amphetamine (oral, 0.5 mg/kg) to measure cortical dopamine transmission in cocaine dependent individuals and healthy controls

DETAILED DESCRIPTION:
This study seeks to examine dopamine (DA) transmission in vivo, using positron emission tomography (PET) with [C-11]FLB 457, in cortical regions of interest in subjects who have a history of cocaine dependence. We hypothesize that cocaine dependence is associated with decreases in dopamine in the prefrontal cortical regions compared to controls. This may explain the impulsivity and cognitive deficits that underlie relapse in this disorder.

ELIGIBILITY:
Subjects with Cocaine Dependence INCLUSION CRITERIA

1. Males or Females 18-40
2. Fulfill Diagnostic and Statistical Manual (DSM-IV) Diagnosis for Cocaine Dependence
3. Medically Healthy MAJOR EXCLUSIONS

1. Major medical, psychiatric, co-morbid drug & alcohol use disorders 2. Pregnancy or lactation, 3. Contraindications to MRI 4. Currently employed as radiation worker; or participation in radioactive drug research protocols within the previous year 5. Family History of a psychotic illness or manic episode in first-degree relatives

Healthy Subjects INCLUSION CRITERIA

1. Males or Females 18-40
2. Absence of present or past psychiatric conditions (including alcohol or drug dependence)
3. A negative urine drug screen
4. Medically Healthy

MAJOR EXCLUSIONS

1. Any medical, psychiatric, co-morbid drug & alcohol use disorders
2. Pregnancy or lactation,
3. Contraindications to MRI
4. Currently employed as radiation worker; or participation in radioactive drug research protocols within the previous year
5. Family History of a psychotic illness or manic episode, or drug and alcohol Abuse/Dependence in first-degree relatives

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-06-02 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Percent change in Binding potential (BPnd) | Baseline BPnd (time 0) and Post-amphetamine BPnd (time 3 hours)
  DELTA BPnd

CONTACTS AND LOCATIONS:
Locations (1):
- University of PIttsburgh PET Facility, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No